CLINICAL TRIAL: NCT03854552
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 764198 in Healthy Male Subjects (Single-blind, Partially Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study in Healthy Men Tests How Different Doses of BI 764198 Are Taken up in the Body and How Well They Are Tolerated.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1434-0001; 2018-004432-30 (EudraCT Number)
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 764198 (Experimental): Single rising oral doses
  Interventions: Drug: BI 764198
- Placebo (Placebo Comparator): Single rising oral doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 764198 — capsule
  Arms: BI 764198
Drug: Placebo — capsule
  Arms: Placebo

SUMMARY:
The main objective of this trial is to investigate safety and tolerability of BI 764198 in healthy male subjects following oral administration of single rising doses.

Secondary objectives are the exploration of pharmacokinetics (PK) including dose proportionality of BI 764198 after single oral dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects who meet any of the following criteria from administration of trial medication until 30 days after trial completion:

  * Males who are willing to use a medically acceptable method of contraception. Acceptable methods of contraception for use by male subjects include sexual abstinence, a vasectomy performed at least 1 year prior to dosing, and barrier contraception (condom)
  * Subjects who are not vasectomised or sexually abstinent have to ensure that an additional acceptable method of contraception will be used by his female partner such as intrauterine device (IUD), surgical sterilisation (including hysterectomy), hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to drug administration, or barrier method (e.g. diaphragm with spermicide)

Exclusion criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance; Creatinine, LFTs (ALT, AST, bilirubin [not exclusionary in subjects with known Gilbert's disease]) and platelets strictly below upper limit of reference range, eGFR strictly ≥ 90 ml/min/1,73 m² (based on CKD-EPI formula)
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 24 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Detection of cataract in slit lamp examination.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with drug-related adverse events (AEs) | From drug administration till the end of trial, up to 14 days.
  The percentage of subjects with drug-related adverse events (AEs).

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 764198 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Within 2 hours (h) prior and 30 minutes (min), 1h, 1h and 30min, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 72h, 96h, 120h and 168h following drug administration.
  Area under the concentration-time curve of BI 764198 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Maximum measured concentration of BI 764198 in plasma (Cmax) | Within 2 hours (h) prior and 30 minutes (min), 1h, 1h and 30min, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 72h, 96h, 120h and 168h following drug administration.
  Maximum measured concentration of BI 764198 in plasma (Cmax).

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Schultz A, Halabi A, Seitz F, Lemmens K, Wulfrath HS, Lobmeyer MT, Retlich S, Choi W, Soleymanlou N. Phase 1 trials of BI 764198, a transient receptor potential channel 6 inhibitor, in healthy volunteers and participants with kidney impairment. Expert Opin Investig Drugs. 2025 May;34(5):415-423. doi: 10.1080/13543784.2025.2510673. Epub 2025 Jun 8. PMID 40455255
- See also: Related Info — https://trials.boehringer-ingelheim.com/